CLINICAL TRIAL: NCT05188352
Title: Effects of Supervised Aerobic Exercise Training on Respiratory Parameters, Exercise Capacity, and Anxiety in Patients With Coronary Artery Bypass Surgery
Brief Title: Exercise Training in Patients After Bypass Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BVUsozyilmaz09
Record Dates: First submitted 2021-12-27; First posted 2022-01-12 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-12

CONDITIONS: Coronary Artery Bypass Surgery
Keywords: coronary artery patients; coronary artery bypass surgery; respiratory muscle strength; oxygen consumption; aerobic exercise; pulmonary function test; maximal exercise test with oxygen consumption

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training group (Experimental): Patients in the training group received supervised aerobic exercise training on the treadmill with the intensity of 60-75% of maximal VO2 for 40-50 minutes, 3 days a week for 8 weeks. Work-load was gradually increased during the eight-week period. In addition, conventional chest physiotherapy and was instructed to continue their daily physical activity program at home patients in this group.
  Interventions: Other: Chest physiotherapy; Other: Aerobic exercise training
- Control group (Active Comparator): Patients in the control group received no aerobic exercise training but were asked to continue their chest physiotherapy and daily physical activity program at home.
  Interventions: Other: Chest physiotherapy

INTERVENTIONS:
Other: Chest physiotherapy — The program included diaphragmatic breathing exercises, thoracic expansion exercises, incentive spirometer exercises, and coughing techniques.
Other: Aerobic exercise training — A treadmill was used for aerobic exercise. Training intensity was used at 60-75% of maximal VO2.
  Each session had a five-minute warm-up and cool-down period. Blood pressure and ECG were recorded during training sessions before exercise, at the third minute of each workload, after exercise, and during each minute of the recovery period.
  Arms: Training group

SUMMARY:
Based on clinical experience both physical condition and psychological recovery after surgery are individually variable. Exercise training plays an important part, has been recommended for CABS patients in order to enhance recovery. Regular exercise following CABS has shown that, in addition to the expected improvements in exercise capacity as a result of the surgery itself, patients who participate in cardiac rehabilitation can expect to see additional gains in exercise capacity and risk factor profiles. Exercise training also increases personal self-esteem and self-confidence, can alleviate depression and fear, and increase the sense of well-being. The aim of this study was to examine the effects of supervised aerobic exercise training on pulmonary function, functional capacity, maximal exercise capacity, and anxiety in patients after coronary artery bypass surgery.

DETAILED DESCRIPTION:
Patients in the training group received supervised aerobic exercise training on the treadmill with the intensity of 60-75% of maximal VO2 for 40-50 minutes, 3 days a week for 8 weeks in a cardiac rehabilitation unit. Work-load was gradually increased during eight-week period. Each session had a five-minute warm-up and cool-down period. Blood pressure and ECG were recorded during training sessions before exercise, at the third minute of each workload, after exercise, and during each minute of the recovery period. In addition, conventional chest physiotherapy and was instructed to continue their daily physical activity program at home patients in this group Patients in the control group received no aerobic exercise training but were asked to continue their chest physiotherapy and daily physical activity program at home.

The same researcher, who was blind to the group allocation, were evaluated all patients for pulmonary functions, respiratory muscle strength and submaximal functional capacity, exercise capacity, and anxiety level initially and after 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male gender,
* CABG surgery performed in the last one month,
* Patients with negative exercise test (on the 30 days after discharge).

Exclusion Criteria:

* Valve surgery,
* Perioperative myocardial infarction assessed by electrocardiographic (ECG) and creatine kinase isoenzyme changes,
* Postoperative angina, diabetes mellitus, chronic renal failure, unstable angina, intermittent claudication, heart valve dysfunction (moderate or severe), severe cardiac arrhythmias, -Presence of symptoms at rest or with minimal exertion,
* Chronic obstructive pulmonary disease (>70% FEV1/FVC), and
* Any disorder that might influence exercise performance physically (e.g. severe back pain, history stroke).

Ages: 35 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline maximum inspiratory pressure at 8 weeks. | [ Time Frame: Eight weeks ]
  Change from baseline Maximum Inspiratory Pressure (MIP) at 8 weeks. Respiratory muscle strength was measured according to the portable, electronic intraoral pressure measuring device (MicroRPM, Micro Medical UK), American Thoracic Society (ATS) and European Respiratory Society (ERS) criteria. The most commonly used method for evaluating respiratory muscles is MIP measurement is a non-invasive technique.
Change from baseline maximum expiratory pressure at 8 weeks | [ Time Frame: Eight weeks ]
  Change from baseline Maximum Expiratory Pressure (MEP) at 8 weeks. Respiratory muscle strength was measured according to the portable, electronic intraoral pressure measuring device (MicroRPM, Micro Medical UK), American Thoracic Society (ATS) and European Respiratory Society (ERS) criteria. The most commonly used method for evaluating respiratory muscles is MEP measurement is a non-invasive technique.
Maximal exercise capacity | [ Time Frame: Eight weeks ]
  The incremantal, symptom-limited cardiopulmonary exercise test (CPET) was used to assess exercise capacity.
  Symptom-limited maximal exercise test with oxygen consumption measurement (peak VO2) (Minjhard Oxycon-3) on the treadmill using a Modified Bruce protocol.

SECONDARY OUTCOMES:
Change from baseline distance covered in six-minute walk test at 8 weeks. | [ Time Frame: Eight weeks ]
  Change from baseline functional capacity test at 8 weeks. Functional capacity was assessed by the 6 minute walking test. The test was performed according to American Thoracic Society (ATS) criteria. Patients were allowed to rest for 10 minutes before the test. Heart rate, blood pressure, respiratory frequency, oxygen saturation, fatigue and dyspnea perception were recorded before and after the test. Walking distance was calculated.
Change from baseline Forced Vital Capacity (FVC) at 8 weeks | [ Time Frame: Eight weeks ]
  Change from baseline Forced Vital Capacity (FVC) in respiratory function test at 8 weeks. FVC was evaluated using spirometry, according to the American Thoracic Society (ATS) and European Respiratory Society (ERS) criteria.
Change from baseline Forced Expiratory Volume in 1 second (FEV1) at 8 weeks . | [ Time Frame: Eight weeks ]
  Change from baseline Forced Expiratory Volume 1 second (FEV1) in respiratory function at 8 weeks. FEV1 was evaluated using spirometry, according to the American Thoracic Society (ATS) and European Respiratory Society (ERS) criteria.
Change from baseline Forced Expiratory flow from between 25% to 75% of Vital Capacity at 8 weeks. | [ Time Frame: Eight weeks ]
  Change from baseline Forced Expiratory flow from between 25% to 75% of Vital Capacity at 8 weeks.
  FMF was evaluated using spirometry, according to the American Thoracic Society (ATS) and European Respiratory Society (ERS) criteria.
Change from baseline anxiety level at 8 weeks. | [ Time Frame: Eight weeks ]
  Anxiety level was evaluated by STAI-I and II.
Change from baseline maximal oxygen consumption(VO2max) level at 8 weeks | [ Time Frame: Eight weeks ]
  Respiratory parameters were continuously measured by using computerized 'Minjhard Oxycon-3'. Measurements were performed in each 30 second, before, during and after exercise test and during each recovery period for five minutes parameters measured.
Change from baseline maximal respiratory minute volume (VE), level at 8 weeks | [ Time Frame: Eight weeks ]
  Respiratory parameters were continuously measured by using computerized 'Minjhard Oxycon-3'. Measurements were performed in each 30 second, before, during and after exercise test and during each recovery period for five minutes parameters measured
Change from baseline VO2max/kg level at 8 weeks | [ Time Frame: Eight weeks ]
  Respiratory parameters were continuously measured by using computerized 'Minjhard Oxycon-3'. Measurements were performed in each 30 second, before, during and after exercise test and during each recovery period for five minutes parameters measured
Change from baseline maximal oxygen pulse (O2pulse) level at 8 weeks | [ Time Frame: Eight weeks ]
  O2 pulse value was calculated from VO2 value which was divided to (by) heart rate at that minute.
Change from baseline maximal MET level at 8 weeks | [ Time Frame: Eight weeks ]
  Respiratory parameters were continuously measured by using computerized 'Minjhard Oxycon-3'. Measurements were performed in each 30 second, before, during and after exercise test and during each recovery period for five minutes parameters measured

CONTACTS AND LOCATIONS:
Overall Officials: Semiramis Özyılmaz, Assoc. Prof., Study Chair — Bezmialem Vakif University